CLINICAL TRIAL: NCT03050411
Title: A Study of Apatinib Combine With EGFR-TKI for Advanced EGFR-TKI-resistant Non-Small Cell Lung Cancer
Brief Title: Apatinib Combine With EGFR-TKI for Advanced EGFR-TKI-resistant Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Li Liang, Prof. M.D., Peking University Third Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00006761-2016162
Record Dates: First submitted 2017-01-09; First posted 2017-02-10 (Actual); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Nonsmall Cell Lung Cancer
Keywords: Non Small Cell Lung Cancer; EGFR-TKI resistance; Apatinib; anti-angiogenesis drugs
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — apatinib; Erlotinib Hydrochloride; Gefitinib; osimertinib

ARMS (1):
- Apatinib (Experimental): Apatinib in combination with EGFR-TKIs
  Interventions: Drug: Apatinib Mesylate Tablets; Drug: EGFR-TKIs (Erlotinib, Gefitinib and Osimertinib)

INTERVENTIONS:
Drug: Apatinib Mesylate Tablets — 250mg, 500mg, 750mg, q.d., p.o.
Drug: EGFR-TKIs (Erlotinib, Gefitinib and Osimertinib) — EGFR-TKIs include but are not limited erlotinib, gefitinib and osimertinib

SUMMARY:
Epidermal growth factor receptor tyrosine kinase inhibitors (EGFR-TKIs), including gefitinib demonstrate excellent effect on the treatment of non-small cell lung cancer (NSCLC) patients with EGFR mutations. However, patients who are initially sensitive to the drugs eventually become resistance. Apatinib is a highly selective VEGFR2 inhibitor and reduces the angiogenesis of tumor efficiently. In this study, the investigators aim to explore the efficacy and reasonable dosage of apatinib combining with EGFR-TKI in advanced non-squamous non-small cell lung cancer with EGFR-TKI resistance.

DETAILED DESCRIPTION:
Primary Outcome Measure: efficacy and reasonable dosage of the combination of apatinib and EGFR-TKI in advanced non-squamous non-small cell lung cancer with EGFR-TKI resistance.

Secondary Outcome Measures: Progression free survival, overall survival, Side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Obtain of informed consent.
2. Histologically or cytologically confirmed, inoperable, recurrence or metastasis advanced non-small cell lung cancer (TNM Stage ⅢB or stage Ⅳ), took EGFR-TKI longer than 6 months and appeared disease progression.
3. At least one measurable lesion (helical CT scan long diameter ≥10mm, meet the requirements of the standard Response Evaluation Criteria In Solid Tumors（RESCIST） version 1.1).
4. Eastern Cooperative Oncology Group（ECOG）Performance Status（PS） :0-2.
5. Aged from 18 to 75 years (18 and 75 years are included).
6. Life expectancy ≥12 weeks.
7. Adequate bone marrow reserve and organ function as follows:

   * Absolute neutrophils count (ANC) ≥1.5 x 10 to the 9th power/L (band neutrophil and segmented neutrophil), platelets > 100 x 10 to the 9th power/L and Hb≥90g/L.
   * Hepatic: total bilirubin less than or equal to 1.5 times upper limit of normal (ULN).
   * Alkaline phosphatase (AP), alanine transaminase (ALT) and aspartate transaminase (AST) less than or equal to 3.0 times ULN (or less than or equal to 5 times ULN in case of known liver involvement.
   * Renal: Serum Creatinine less than or equal to 1.25 times upper limit of normal (ULN).
8. Have history of hypertension (less than 135/85mmHg).
9. Females of child-bearing potential must have negative serum pregnancy test. Sexually active males and females (of childbearing potential) willing to practice contraception during the study.

Exclusion Criteria:

1. Do not meet the above criteria.
2. Prior treatment with VEGFR tyrosine kinase inhibitors or VEGFR targeting agent.
3. Unhealed toxicity of prior anti-cancer treatment (CTCAE Level 1) or surgery.
4. Symptomatic Central Nervous System (CNS) metastases.
5. Uncontrolled hypertension (systolic ≥140mmHg and/or diastolic ≥90mmHg after medication treatment).
6. Clinical uncontrolled active infection, such as acute pneumonia, active hepatitis B or C (prior hepatitis B history, despite medication treatment control or not, HBV DNA≥500copies or ≥100IU/ml), etc.
7. Arterial thrombosis or venous thrombosis in 6 months, or disposition evidence of thrombosis/bleeding in 2 month (despite severity), hemoptysis in 2 weeks (bright red blood, 1/2 teaspoon).
8. Stroke or transient ischemic attack (TIA) in 12 month.
9. Unhealed skin lesions, surgical site, injuries, severe mucous membrane ulcer or bone fracture.
10. Cardiac function evaluation: LVEF <50%, a recent history of MI in 6 months, severe/unstable angina or coronary bypass surgery, or cardiac insufficiency ≥ NYHA 2.
11. Prior other malignant disease in 5 years (except carcinoma in situ of cervix, or non melanoma skin cancers, or localized prostate cancer with Gleason ≤6).
12. Documented history of neurological or psychiatric disorders, include epilepsy and dementia.
13. Recent active digestive disease such as duodenal ulcers, ulcerative colitis, ileus, ect., intestinal perforation, intestine fistula, or other conditions may lead to gastrointestinal bleeding or perforation which regimented at investigators' discretion.
14. Difficulty swallowing or known malabsorption.
15. A history of organ transplantation and long-term immunosuppressive medication.
16. Take part in new drug clinical trials within one month or taking part in a trial now.
17. Pregnant or lactating woman.
18. A history of anaphylaxis of apatinib analogue and/or excipient of drugs in this study.
19. Other conditions regimented at investigators' discretion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-05; Primary Completion 2019-06 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Optimal Dosage | 9 months
  Optimal dosage of Apatinib which combine with EGFR-TKIs
Progression free survival | 24 months
  PFS is evaluated in 24 months since the treatment begin

SECONDARY OUTCOMES:
Overall survival | 24 months
  Overall survival is evaluated in the 24th month since the treatment began
Side effects | 24 months
  Side effects evaluated in the 24th month since the treatment began according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Li Liang, Prof. M.D., Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China